CLINICAL TRIAL: NCT03554148
Title: Assessment of Bacterial Translocation on the Incidence of Surgical Site Infection in Abdominal Surgery: Prospective Cohort Study.
Brief Title: Bacteria and Intestinal Translocation in Surgery (Bandit)
Acronym: Bandit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: Bandit
Record Dates: First submitted 2017-11-09; First posted 2018-06-12 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SSI: This group receives an additional swab of the surgical site infection. Follow up is terminated at the occurence of SSI.
  Interventions: Other: No intervention
- No SSI: This group is systematically followed up until 30 days after surgery (one year if a implant is implanted, e.g. mesh) by a third party (www.swissnoso.ch).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is purely an observational study. Groups SSI/No SSI are defined by the occurence of a surgical site infection.

SUMMARY:
Patients undergoing elective abdominal surgery will be included prospectively. Informed consent will be obtained. Preoperatively baseline health data is collected and a skin swab and rectal swab for baseline skin and gut microbiota is taken. During the surgery additional clinical data and additional samples will be obtained. Additional samples include: rectal swab, biopsies of the resected specimen (lymph node, peritoneum, intestinal content, mucosa), venous blood sample (7.5ml) at the end of the operation, liver biopsy and skin biopsy. Postoperative health data is recorded. If a surgical site infection occurs a swab is taken too. With 16 sRNA (small ribonucleic acid) based sequencing the investigators will quantify the abundance of the different bacterial species in all samples. Primary outcome will be to assess a difference of 16sRNA signal in the liver and lymph node biopsies between patients with and patients without surgical site infection. Secondary outcomes include variables predicting the occurence of surgical site infections and a model describing the way bacteria may take to cause wound infection.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* All Ages
* All Gender
* Elective Abdominal Surgery
* Age > 18
* All approached (laparoscopic, open)
* All ethnic and sociodemographic backgrounds
* Sufficient knowledge of the study language (German)

Exclusion Criteria:

* pregnant or lactating women
* no operation performed (i.e. only planned)
* insufficient knowledge of project language (German)
* lack of informed consent
* known colonization with multi-resistant bacteria (e.g. Methicillin-resistant Staphylococcus aureus (MRSA) or extended spectrum betalactamase (ESBL))
* known cirrhotic liver disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing elective visceral surgery. Mostly for oncological indications.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of bacterial DNA in liver biopsy | day 0 (operation day)
  Rationale: One of the aims is to test how the liver acts as primary barrier for blood-borne bacteria during the operation.
  Sampling: During elective abdominal surgery a biopsy with the Tru-Cut™ Needle (Baxter healthcare Co., 16G Chicago, USA) is performed as recommended by the manufacturer. Hemostasis is achieved by Application of mono-polar Electrocautery.
  Processing: The sample is immediately snap-frozen in liquid nitrogen. Storage: Biobank: -80°C. Analysis: Polymerase chain reaction (PCR) with bacteria specific primers, Sequencing of the PCR product (IonTorrent) to determine the present microbiota (species if possible, at least families). The difference in positive/negative liver probes is compared for patients with and without surgical site infections (Chi squared Test).

SECONDARY OUTCOMES:
Detection of bacterial DNA in mesenteric lymph node | day 0 (operation day)
  Rationale: To address the interstitial translocation and drainage of microbes during colonic surgery. Positive lymph nodes are a surrogate marker of SSI. However, positive lymph nodes may just be a surrogate a marker of a high amount of bacteria being translocated from intestinal lumen to the interstitial space during surgery. Or, mesenteric lymph nodes truly are a significant line of defence against surgical site infections.
  Sampling: A lymph node is sampled from the resected specimen within the OR under sterile conditions. The lymph node is excised. Half of this lymph node is sampled for research purposes, the other half is marked with a suture and sent for pathological evaluation with the rest of the specimen.
  Processing: Sample is immediately snap-frozen in liquid nitrogen. Storage: Biobank: -80°C. Analysis: same as liver biopsy. The difference in positive/negative lymph node probes is compared for patients with and without surgical site infections (Chi squared Test).
Number of patients with surgical site infection (SSI) | outpatient visit, usually around 7 to 21 days before operation
  The number of patients with surgical site infection are recoded. Surgical site infection is defined according to the Centers for Disease Control and Prevention Guideline for the Prevention of Surgical Site Infection, 2017.
Modelling bacterial travel behaviour in multimodal networks | day 0
  Rationale: The way bacteria travel from places they grow in abundance(gut,skin), ending up in a surgical site to cause infection, has not been studied.
  Sampling: In addition to the preoperative skin and rectal swab and the intraoperative liver and lymph node biopsy, additional samples are collected in a prospective manner: biopsy of the visceral peritoneum, parietal peritoneum, intestinal mucosa and skin. Swab of intestinal content. Venous blood. All samples are handled sterile and are immediately frozen in liquid nitrogen and stored at -80°C.
  Analysis: For the surgical site infections subgroup, samples are analyzed as described above(bacteria specific PCR followed by Sequencing). The sequencing results translate tinto abundance of families/species. Multimodal networks are applied to describe the potential travel behaviour of bacteria.
Baseline skin and gut microbiota | outpatient visit, usually around 7 to 21 days before operation
  The baseline gut and skin microbiota are metagenomically characterized on the basis of 16S rRNA genomic DNA sequencing.
  Statistical analysis: Differences of skin and gut microbiota between patients with and without surgical site infections are compared using PerMANOVA. The correlation between distinct microbiota (families or clusters) and the occurence surgical site infections is tested using multiple logistic regressions.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Beldi, MD, Prof, Study Director — Inselspital, University Hospital of Bern
Locations (1):
- Inselspital, University Hospital Bern, Visceral Surgery Department, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided